CLINICAL TRIAL: NCT05891509
Title: Efficacy and Safety of DTI-guided Minimally Invasive Hematoma Evacuation Versus Best Medical Therapy for Acute Spontaneous Intracerebral Hemorrhage: a Randomized Controlled Trial
Brief Title: DTI-guided Minimally Invasive Hematoma Evacuation for Intracerebral Hemorrhage
Acronym: GLAMOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongming Qiu (Other)
Collaborators: Xingguo County People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Organization: Xinqiao Hospital of Chongqing (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLAMOR
Record Dates: First submitted 2023-05-28; First posted 2023-06-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Stroke Hemorrhagic
Keywords: Minimally Invasive Hematoma Evacuation; Intracerebral Hemorrhage; Randomized Controlled Trial; Magnetic Resonance Imaging
MeSH Terms: conditions — Hemorrhagic Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: Other design features: The investigators will conduct a multicenter randomized controlled trial, as well as a concurrent prospective observational study including all ICH patients who decline participation in the trial and will therefore receive minimally invasive hematoma evacuation or best medical therapy and consent to be followed up. All participants will be followed up at the same time using the same outcomes measures. The primary outcome will be collected by a blinded assessor.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Invasive Hematoma Evacuation (Experimental): Subjects randomized to this arm will receive the intervention of minimally invasive hematoma evacuation and best medical therapy
  Interventions: Procedure: Minimally Invasive Hematoma Evacuation; Other: Best Medical Therapy
- Best Medical Therapy (Active Comparator): Subjects randomized to this arm will receive best medical therapy alone
  Interventions: Other: Best Medical Therapy

INTERVENTIONS:
Procedure: Minimally Invasive Hematoma Evacuation — Procedure of minimally invasive hematoma evacuation PLUS best medical therapy
  Arms: Minimally Invasive Hematoma Evacuation
Other: Best Medical Therapy — Best medical therapy

SUMMARY:
Intracerebral hemorrhage (ICH) is a devastating disease with high early mortality, unfavorable neurological outcomes, and high cost of care. To date, the role of DTI-guided minimally invasive hematoma evacuation in ICH is still uncertain.

The investigators will conduct a multicenter randomized controlled trial, as well as a concurrent prospective observational study including all ICH patients who decline participation in the trial and will therefore receive minimally invasive hematoma evacuation or best medical therapy and consent to be followed up. All participants will be followed up at the same time using the same outcomes measures. The primary outcome will be collected by a blinded assessor.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. Intracerebral hemorrhage in the basal ganglia was diagnosed by CT examination;
3. The amount of bleeding is 20-40ml, and the midline structure is displaced horizontally by < 3mm in the pineal gland;
4. The degree of integrity and continuity of the corticospinal tract on the lesion side of magnetic resonance diffusion tensor imaging was graded as grade 2~4;
5. The time from onset to randomization is within 24 hours;
6. GCS score ≥ 4 points at randomization;
7. Muscle strength level 3 in the affected limb;
8. Written informed consent are provided by the patients or their legal representatives.

Exclusion Criteria:

1. Bleeding in other parts (e.g., bleeding in subtentorial areas such as thalamus, brainstem or cerebellum);
2. Bleeding caused by other causes (such as aneurysm, arteriovenous malformation, brain trauma, brain tumor, bleeding transformation of large cerebral infarction, bleeding caused by β amyloidosis, bleeding caused by coagulation dysfunction) or combined with aneurysm, arteriovenous malformation, brain trauma, brain tumor, large-scale cerebral infarction, β amyloidosis, severe coagulation dysfunction;
3. Multiple intracranial hemorrhage;
4. Patients with ventricular hemorrhage or ICH rupture into the ventricles should consider the need for ventricular drainage;
5. Any history of brain parenchymal or other intracranial subarachnoid, subdural or epidural hemorrhage and surgical history in the past 30 days;
6. Myocardial infarction within the past 30 days;
7. Previous history of bleeding, such as gastrointestinal bleeding, genitourinary bleeding, respiratory bleeding that has not been completely controlled;
8. Hemoglobin < 100g/L, hematocrit <25%, platelet count < 100*109/L;
9. Receiving anticoagulant drugs such as warfarin, dabigatran or rivaroxaban within 1 week prior to enrollment, with an INR > 1.4;
10. Long-term anticoagulation and antiplatelet therapy are expected to be required;
11. Allergy to alpeplase, urokinase or surgery-related drugs and instruments;
12. Pregnant or lactating women;
13. Known high risk of embolism, including patients with mechanical heart valves implanted in the body, history of left heart thrombosis, mitral stenosis with atrial fibrillation, acute pericarditis, or subacute bacterial endocarditis. Atrial fibrillation without mitral stenosis is appropriate;
14. hypertension (systolic blood pressure is still greater than 180mmHg) that cannot be effectively controlled by aggressive antihypertensive therapy before randomization;
15. Life expectancy < 12 months in the advanced stage of any disease;
16. Participating in other interventional clinical studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of score of 0-3 on the modified Rankin scale | 180 days after randomization
  Scores on the modified Rankin scale range from 0 to 6, with higher scores indicating greater disability.

SECONDARY OUTCOMES:
Score of on the modified Rankin scale | 180 days after randomization
  Scores on the modified Rankin scale range from 0 to 6, with higher scores indicating greater disability.

OTHER OUTCOMES:
Incidence of symptomatic intracranial hemorrhage | 30 days after randomization
  Symptomatic intracranial hemorrhage will be defined according the Heidelberg bleeding classification criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Xingguo County People's Hospital, Ganzhou, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code